CLINICAL TRIAL: NCT04993157
Title: A Phase I, Single-dose, Open-label, Parallel-group Study to Assess the Pharmacokinetics, Safety, and Tolerability of FIA586 in Participants With Mild and Moderate Hepatic Impairment Compared to Matched Healthy Participants
Brief Title: Pharmacokinetics Study of FIA586 in Participants With Mild and Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFIA586A02101
Record Dates: First submitted 2021-08-03; First posted 2021-08-06 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; NASH; Child-Pugh classification; FIA586

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Healthy participants with normal hepatic function (Experimental): Each participant will receive a single dose of FIA586
  Interventions: Drug: FIA586
- Group 2: Participants with mild hepatic impairment (Experimental): Each participant will receive a single dose of FIA586
  Interventions: Drug: FIA586
- Group 3: Participants with moderate hepatic impairment (Experimental): Each participant will receive a single dose of FIA586
  Interventions: Drug: FIA586

INTERVENTIONS:
Drug: FIA586 — FIA586 capsule

SUMMARY:
This is a Phase I study designed to characterize the pharmacokinetics (PK), safety, and tolerability of a single oral dose of FIA586 in participants with mild and moderate hepatic impairment (HI) compared to matched healthy participants.The information obtained in this study will help to determine whether dosage adjustment for FIA586 is necessary in patients with advanced liver fibrosis who have mild to moderate HI.

DETAILED DESCRIPTION:
This is a Phase I, single-dose, open-label, parallel-group study in participants with mild (Child-Pugh A; n=8-10) and moderate (Child-Pugh B; n=8-10) hepatic impairment (HI) and matched healthy participants with normal hepatic function (n=8-20).

The study is comprised of an up to 28-day screening period (Days -28 to 2), a baseline evaluation (Day -1) prior to dosing on Day 1, and a treatment period of 6 days (Days 1-6). Participants will remain domiciled up to Day 6 after the Study Completion procedures have been completed.

On Day 1, participants will be given a single dose of FIA586 following an overnight fast. PK (plasma and urine) and biomarker samples will be taken prior to dosing of study treatment and up to 120 hours (Day 6) post- dose. On Day 6, after the last PK sample has been taken, Study Completion assessments will be performed, and the participant will be discharged, provided there are no safety or tolerability concerns as judged by the investigator.

All participants will have a post-study safety contact conducted approximately 30 days after administration of study treatment.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Male and non-childbearing potential female participants 18 to 70 years of age (inclusive) at Screening.
* Must weigh at least 50.0 kg and must have a body mass index (BMI) within the range of 18.0 to - 38.0 kg/m2 at Screening.
* Must be a non-smoker or agree to smoke no more than 5 cigarettes (or equivalent) per day, and maintain the same smoking status from Screening until the Study Completion (Day -28 to Day 6).

Healthy participants (Group 1)

* Must be in good health as determined by past medical history, physical examination, vital signs, ECG, and laboratory tests at Screening.
* Each participant must match in age (±10 years), gender, weight (±15%), and smoking status (smoker or non-smoker) to an individual participant in at least one HI group but not to more than 1 participant in the same HI group.

Participants with mild and moderate HI (Groups 2 and 3)

• Must satisfy the criteria for HI as evidenced by a Child-Pugh class of A or B at Screening:

* Class A; Mild; Child-Pugh score 5-6
* Class B; Moderate; Child-Pugh score 7-9

Exclusion Criteria:

All participants:

* Use of other investigational drugs within the last 30 days or 5 half-lives prior to dosing of study treatment, whichever is longer.
* Known history of, or current clinically significant arrhythmias. Have clinically significant ECG abnormality or history of long-QT syndrome.
* Myocardial infarction < 5 years prior to Screening.
* Recent (within the last 3 years of Screening) or recurrent history of autonomic dysfunction (e.g. recurrent episodes of fainting or palpitations).
* History of immunodeficiency diseases or have a positive HIV test result at Screening.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 3 years of Screening, regardless of whether there is evidence of local recurrence or metastases.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs (apart from cholecystectomy), or which may jeopardize the participants in case of participation in the study. The investigator should make this determination in consideration of the participant's medical history and/or clinical or laboratory evidence of any of the following:

  * Inflammatory bowel disease, peptic ulcers, gastrointestinal including rectal bleeding within 3 months prior to Screening.
  * Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection.
  * Pancreatic injury or pancreatitis.

Healthy participants (Group 1):

* Any single parameter of alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transferase (GGT), or alkaline phosphatase (ALP) exceeding 1.2 × upper limit of normal (ULN) or ≥ 1.5 × ULN total bilirubin (TBL) OR any elevation above ULN of more than one parameter of ALT, AST, GGT, ALP, or serum bilirubin at screening.
* Known to have Gilbert's syndrome.
* Hemoglobin levels below 12.0 g/dL for males and 11.0 g/dL for females at Screening or Baseline.
* History or presence of impaired renal function as indicated by clinically significant abnormal creatinine or blood urea nitrogen (BUN) and/or urea values, or abnormal urinary constituents at Screening.
* Total white blood cell (WBC) count which falls outside the range of 3.5 to 10.7 × 109/L, or platelets < 100 × 109/L at Screening or Baseline.
* Evidence of urinary obstruction or difficulty in voiding at Screening.
* Symptomatic genital or urinary tract infection in the 4 weeks prior to dosing of study treatment or the presence of active urinary tract infection at Screening.

Participants with mild and moderate HI (Groups 2 and 3):

* Have abnormal laboratory values for any of the following parameters at Screening or Baseline:

  * Hemoglobin < 9 g/dL.
  * Platelet count < 30 × 109/L.
  * WBC count < 2.5 × 109/L.
  * Absolute neutrophil count < 1.5 × 109/L.
  * Lymphocytes < 0.8 × 109/L.
  * TBL > 8 mg/dL.
  * Serum amylase > 2 × ULN.
  * International normalized ratio (INR) > 2.3
  * Corrected serum calcium < 8.6 or > 10.2 mg/dL.
* Hepatic impairment due to non-liver disease.
* Presence of any non-controlled and clinically significant disease that could affect the study outcome or that would place the participant at undue risk.
* Treatment with any vasodilator, autonomic alpha blocker or β2 agonist within 2 weeks prior to dosing of study treatment.
* Primary biliary cholangitis or biliary obstruction.
* Participants requiring paracentesis more than every 30 days for the management of ascites are excluded. Participants who are receiving diuretics to manage ascites may be enrolled and will be assigned the Child-Pugh score for the degree of ascites while on diuretic treatment. The diuretic dose must have been stable for 28 days prior to dosing of study treatment.
* Have transjugular intrahepatic portosystemic shunt and/or have undergone portacaval shunting.
* Have encephalopathy Grade 3 or worse within 28 days prior to dosing of study treatment.
* Presence of moderate to severe impaired renal function as indicated by estimated glomerular filtration rate (eGFR) < 50 mL/min/1.73 m2 based on the modification of diet in renal disease calculation at Screening.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Blood Concentrations (Cmax) for FIA586 | pre-dose, 0.25 hours, 0.5 hours, 1 hour, 1,5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours, 72 hours, 92 hours and 120 hours
  Blood samples will be collected to measure Cmax at indicated time-points. Pharmacokinetic (PK) parameters will be calculated based on FIA586 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC MS/MS) method with a lower limit of quantification of 20 ng/mL. Cmax will be determined using non-compartmental methods.
Area Under Plasma Concentration-time Curve from time zero to the last measurable concentration sampling time (AUClast) for FIA586 | pre-dose, 0.25 hours, 0.5 hours, 1 hour, 1,5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours, 72 hours, 92 hours and 120 hours
  Blood samples will be collected to measure AUClast at indicated time-points. Pharmacokinetic (PK) parameters will be calculated based on FIA586 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC MS/MS) method with a lower limit of quantification of 20 ng/mL. AUClast will be determined using non-compartmental methods.
Area Under Plasma Concentration-time Curve from Time Zero Extrapolated to Infinity (AUC[0-inf]) for FIA586 | pre-dose, 0.25 hours, 0.5 hours, 1 hour, 1,5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours, 72 hours, 92 hours and 120 hours
  Blood samples will be collected to measure AUC(0-t) at indicated time-points. Pharmacokinetic (PK) parameters will be calculated based on FIA586 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC MS/MS) method with a lower limit of quantification of 20 ng/mL. AUC[0-inf] will be determined using non-compartmental methods
Area Under Plasma Concentration-time Curve from time 0 to 48 hours (AUC0-48h) for FIA586 | pre-dose, 0.25 hours, 0.5 hours, 1 hour, 1,5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours and 48 hours
  Blood samples will be collected to measure AUC0-48h at indicated time-points. Pharmacokinetic (PK) parameters will be calculated based on FIA586 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC MS/MS) method with a lower limit of quantification of 20 ng/mL. AUC0-48h will be determined using non-compartmental methods.
Time to Reach Maximum Blood Concentrations (Tmax) for FIA586 | pre-dose, 0.25 hours, 0.5 hours, 1 hour, 1,5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours, 72 hours, 92 hours and 120 hours
  Blood samples will be collected to measure Tmax at indicated time-points. Pharmacokinetic (PK) parameters will be calculated based on FIA586 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC MS/MS) method with a lower limit of quantification of 20 ng/mL. Tmax will be determined using non-compartmental methods.
Terminal Elimination Half-life (T1/2) for FIA586 | pre-dose, 0.25 hours, 0.5 hours, 1 hour, 1,5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours, 72 hours, 92 hours and 120 hours
  Blood samples will be collected to measure T1/2 at indicated time-points. Pharmacokinetic (PK) parameters will be calculated based on FIA586 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC MS/MS) method with a lower limit of quantification of 20 ng/mL. T1/2 will be determined using non-compartmental methods.
Apparent Clearance (CL/F) of FIA586 | pre-dose, 0.25 hours, 0.5 hours, 1 hour, 1,5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours, 72 hours, 92 hours and 120 hours
  Blood samples will be collected to estimate CL/F at indicated time-points. Pharmacokinetic (PK) parameters will be calculated based on FIA586 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC MS/MS) method with a lower limit of quantification of 20 ng/mL.
Apparent volume of distribution during terminal elimination phase (Vz/F) of FIA586 | pre-dose, 0.25 hours, 0.5 hours, 1 hour, 1,5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 60 hours, 72 hours, 92 hours and 120 hours
  Blood samples will be collected to estimate Vz/F at indicated time-points. Pharmacokinetic (PK) parameters will be calculated based on FIA586 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC MS/MS) method with a lower limit of quantification of 20 ng/mL.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Novartis Investigative Site, Coral Gables, Florida
  - Novartis Investigative Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CFIA586A02101 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18062
- See also: Plain Lanuguage Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1548